CLINICAL TRIAL: NCT02030977
Title: The Effects of Resveratrol Supplement on Lipid Profile, Liver Enzymes, Inflammatory Factors and Hepatic Fibrosis in Patients With Nonalcoholic Steatohepatitis
Brief Title: The Effects of Resveratrol Supplement on Biochemical Factors and Hepatic Fibrosis in Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr Azita Hekmatdoost (Other)
Responsible Party: Sponsor-Investigator, Dr Azita Hekmatdoost, PI, National Nutrition and Food Technology Institute
Organization: National Nutrition and Food Technology Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 046468
Record Dates: First submitted 2013-12-29; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Non Alcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Resveratrol (Active Comparator): Active Comparator: Resveratrol
  1 Resveratrol capsules for 12 weeks
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): one capsule per day
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol
  Other Names: Dietary Supplement: Resveratrol; 1 Resveratrol capsule per day for 12 weeks
  Arms: Resveratrol
Other: placebo
  Arms: Placebo

SUMMARY:
To study the effects of Resveratrol supplement on lipid profile, liver enzymes, inflammatory factors and hepatic fibrosis in patients with Nonalcoholic Fatty Liver (NAfLD), 50 patients who referred to Gastrointestinal (GI) clinic with steatosis grade 1 or more will be randomly allocated to receive 1 Resveratrol capsules or placebos for 12 weeks; both groups will be advised to adherence our diet and exercise program too. At the first and the end of the intervention, lipid profiles, liver enzymes, some inflammatory cytokines, and liver fibrosis will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older;
* Evidence of nonalcoholic steatohepatitis with steatosis grade higher or equal to 1 in ultrasonography;
* No history of Alcohol consumption or consuming less than 10 grams alcohol per day in women and less than 20 grams per day in men;
* Absence of other liver disorders, malignancies, cardiovascular, respiratory, and kidney disorders;
* Absence of pregnancy or lactation;
* Absence of taking any medications in the past three months;
* Absence of weight loss in the recent three months;
* Absence of endocrine and metabolism disorders.

Exclusion Criteria:

* Weight loss more than 10% of baseline body weight during the intervention period.
* Pregnancy;
* Disliking to continue the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Alaninaminotransferase(ALT) | 12 weeks

REFERENCES:
- [Derived] Faghihzadeh F, Adibi P, Rafiei R, Hekmatdoost A. Resveratrol supplementation improves inflammatory biomarkers in patients with nonalcoholic fatty liver disease. Nutr Res. 2014 Oct;34(10):837-43. doi: 10.1016/j.nutres.2014.09.005. Epub 2014 Sep 23. PMID 25311610